CLINICAL TRIAL: NCT02886949
Title: The Relationship of Vascular Cell Adhesion Molecule 1, C-reactive Protein, Brain-derived Neurotrophic Factor, Orexin and Depressive Symptoms in the Subjects With Thyroid Disease
Brief Title: The Association Between Autoimmune or Inflammation and Thyroid Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CE11307
Record Dates: First submitted 2015-09-02; First posted 2016-09-01 (Estimated); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: THYROTOXICOSIS
MeSH Terms: conditions — Thyrotoxicosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples and urine samples
Oversight: Data Monitoring Committee: No

SUMMARY:
This study aims to evaluate the effects of thyroid functions on energy homeostasis and inflammation.

DETAILED DESCRIPTION:
The subjects were enrolled for evaluation of thyroid functions. The associations between thyroid function and energy homeostasis and inflammation will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Subjects visits outpatient department due to a suspicion of thyroid disease

Exclusion Criteria:

* Psychological disorders, severe inflammatory or infection diseases.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with a suspicion of thyroid disease.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2011-11; Primary Completion 2020-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
brain-derived neurotrophic factor | 3 months
  BDNF

SECONDARY OUTCOMES:
vascular cell adhesion molecule 1 (VCAM-1) | 3 months
  Inflammation
C-reactive protein (CRP) | 3 months
  Inflammation
Orexin | 3 month
  Psychological assessment
Zung Self-Rating Depression Scale (Zung SDS) | 3 month
  Depressive symptom
Body composition | 3 month
  fat component
ankle brachial index (ABI) | 3 months
  Arterial stiffness
pulse wave velocity (PWV) | 3 months
  Arterial stiffness
mean arterial pressure (MAP) | 3 months
  Arterial stiffness

CONTACTS AND LOCATIONS:
Overall Officials: I-Te Lee, MD, Principal Investigator — Taichung Veterans General Hospital
Locations (1):
- Division of Endocrinology and Metabolism, Department of Internal Medicine, Taichung Veterans General Hospital, Taichang, Taiwan

IPD SHARING:
Plan to Share IPD: No